CLINICAL TRIAL: NCT01925404
Title: Promoting Physical Activity In High Poverty Neighborhoods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: City of Los Angeles Department of Recreation and Parks (Unknown); AltaMed Health Services Corporation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2011-0692-AM02; R01HL114283 (NIH)
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Physical Activity
Keywords: Physical activity; parks; programming; public health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Frequent User Arm (Experimental): Park users will be able to earn rewards or prizes by coming more frequently to the park
  Interventions: Behavioral: Frequent User
- Free Physical Activity Classes/programs (Experimental): We will offer at least 100 free physical activity classes at the park
  Interventions: Behavioral: Free physical activity classes
- Combined arm (Experimental): We will offer free classes and the frequent user program at the park
  Interventions: Behavioral: Free physical activity classes; Behavioral: Frequent User
- Control (No Intervention): Business as usual, no special physical activity programs offered

INTERVENTIONS:
Behavioral: Free physical activity classes — 100 hours of free activity classes will be provided
  Arms: Combined arm; Free Physical Activity Classes/programs
Behavioral: Frequent User — Participants can become eligible for prizes by visiting the park more frequently
  Arms: Combined arm; Frequent User Arm

SUMMARY:
Encouraging greater levels of physical activity is critical to improving health among Americans, who are largely sedentary. Neighborhood parks are resources for physical activity that are available to most Americans within a couple miles of their homes, yet many residents are unaware of the programs and facilities available. Previous research indicates that park use is related to park programming and outreach. Because funding for parks is limited, low-cost interventions are needed to attract more people to parks to engage in moderate-to-vigorous physical activity. While many community-based organizations would like to invest in efforts that increase physical activity, few low-cost park programs are documented to be both scalable and cost-effective. Effective programs that can be replicated to make population-level impacts are needed. The goal of this study is to develop and test 2 low-cost community-level approaches, free exercise classes vs. a frequent user program, to promoting physical activity, singly and in combination, in 48 park settings in Los Angeles low-income neighborhoods.

DETAILED DESCRIPTION:
While routine physical activity is critical to optimal health, our preliminary studies have indicated that residents of low-income communities in Los Angeles are less likely to exercise than those in high-income communities, and they are less likely to use their neighborhood parks, even when the parks are within walking distance. Parks in low-income neighborhoods tend to be smaller and serve a greater population density, but even after accounting for the size and the population served, they are still used less than parks in wealthier neighborhoods. In our preliminary studies we found that parks in low-income neighborhoods also had fewer part-time staff and offered fewer programs and organized activities than parks in higher-income areas, and these factors partly accounted for their lower use. As well, parks in low-income neighborhoods are often perceived as less safe, a characteristic associated with lower use 4. Simultaneously, the lack of use and dearth of programming may contribute to a perception of lack of safety, creating a vicious cycle. Nonetheless, we have documented that when parks in low-income neighborhoods offer events and activities, they can be just as busy as parks in higher-income areas. We hypothesize that limited park use in low-income areas can be attributed to the lack of organized and reliable infrastructure of activities that meet the needs of local residents and that offering more activities and programs in parks will increase park use and park-based physical activity.

According to the Task Force on Community Level Preventive Services, community-level campaigns are both effective and scalable.6 For the past eight years, we have conducted research in public neighborhood parks and found that these venues offer great potential for increasing physical activity for populations. Based upon this work, as well as our previous work on the cost-effectiveness of physical activity interventions, we propose to test community-level campaigns targeting low-income populations that will be relatively low-cost and easy to replicate.

The proposed study has three specific aims:

1. Using a full factorial design, compare whether park use and population physical activity in low-income neighborhoods increase with the availability of a) more organized physical activity classes, including zumba, line dancing, and aerobics indoors and outdoors, and/or b) a loyalty program approach that rewards frequent park users.
2. Determine whether either of these two approaches changes the perception of park safety and neighborhood safety.
3. Identify the cost effectiveness of both approaches in terms of dollars spent to generate increased physical activity in parks as measured through systematic observation.

Most Los Angeles parks have full-time staff, but their role has become increasingly administrative. Park staff may not have the time or the skills to lead physical activity programs and activities nor conduct effective outreach to the community to promote these activities. Although there is a small literature on "best practices" for parks, there is no underlying foundation of rigorous scientific research, and there has been no identification of which park practices, designs, or activities lead to the most physical activity in a community. Standard practice is currently based primarily on anecdotes, demands of special interest groups, and the experience of professionals. The science of objectively measuring physical activity in parks is new, developed only in the past decade. Because neighborhood parks are settings designed for moderate to vigorous physical activity (MVPA) and are accessible to 70% of the US population, identifying which programs help populations achieve physical activity goals at a reasonable cost would be highly useful, particularly for groups disproportionately affected with chronic diseases that could be reduced with physical activity. Parks are community resources typically funded by dedicated revenue streams and fee-based programs, yet park systems frequently lack the tools and resources to either market programs or measure their reach or effectiveness. Our study will document all the steps required for implementing and maintaining two physical activity promotion interventions--one a standard approach offering traditional organized physical activity programs, the other an innovative application of popular customer loyalty programs. We will determine their impact on physical activity and their cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria: Parks are in low-income neighborhoods; individuals visit parks and/or live within 1 mile radius of the park; -

Exclusion Criteria: Parks are not in low income neighborhoods; individuals do not visit the park and do not live within a 1 mile radius

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Cohen, MD, MPH, Principal Investigator — RAND
Locations (1):
- RAND, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Yes
May be available upon request as appropriate. We have response data from park users and residents living within one mile of enrolled parks. Interested researchers should contact the PI

REFERENCES:
- [Derived] Derose KP, Han B, Park S, Williamson S, Cohen DA. The mediating role of perceived crime in gender and built environment associations with park use and park-based physical activity among park users in high poverty neighborhoods. Prev Med. 2019 Dec;129:105846. doi: 10.1016/j.ypmed.2019.105846. Epub 2019 Sep 10. PMID 31518627
- [Derived] Cohen DA, Han B, Park S, Williamson S, Derose KP. Park Use and Park-Based Physical Activity in Low-Income Neighborhoods. J Aging Phys Act. 2019 Jun 1;27(3):334-342. doi: 10.1123/japa.2018-0032. Epub 2018 Nov 21. PMID 30160585
- [Derived] Han B, Cohen DA, Derose KP, Li J, Williamson S. Violent Crime and Park Use in Low-Income Urban Neighborhoods. Am J Prev Med. 2018 Mar;54(3):352-358. doi: 10.1016/j.amepre.2017.10.025. Epub 2018 Jan 12. PMID 29338953
- [Derived] Derose KP, Han B, Williamson S, Cohen DA. Gender Disparities in Park Use and Physical Activity among Residents of High-Poverty Neighborhoods in Los Angeles. Womens Health Issues. 2018 Jan-Feb;28(1):6-13. doi: 10.1016/j.whi.2017.11.003. Epub 2017 Dec 11. PMID 29241943

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parks are the unit of analysis; Parks were randomly assigned to the study arms
Units Other Than Participants: Parks
Period: Overall Study
Arm/Group | Frequent User Arm | Free Physical Activity Classes/Programs | Combined Arm | Control
Started (The numbers reported are the number of parks assigned to the study arm) | NA; 12 Parks (The primary outcome of this study is at the level of a park. The park is the unit of analysis. We did not recruit participants, but had measure of park use by counting observed users) | NA; 12 Parks (The park is the unit of analysis. We did not recruit participants, but had measure of park use by counting observed users) | NA; 12 Parks (The park is the unit of analysis. We did not recruit participants, but had measure of park use by counting observed users) | NA; 12 Parks (The park is the unit of analysis. We did not recruit participants, but had measure of park use by counting observed users)
Completed | NA; 12 Parks (We did not recruit participants or follow the same park users over time. The follow up numbers of users are greater than at baseline, and this generates an error message.) | NA; 12 Parks (We did not recruit participants or follow the same park users over time. The follow up numbers of users are greater than at baseline, and this generates an error message.) | NA; 12 Parks (We did not recruit participants or follow the same park users over time. The follow up numbers of users are greater than at baseline, and this generates an error message.) | NA; 12 Parks (We did not recruit participants or follow the same park users over time. The follow up numbers of users are greater than at baseline, and this generates an error message.)
Not Completed | NA; 0 Parks | NA; 0 Parks | NA; 0 Parks | NA; 0 Parks

BASELINE CHARACTERISTICS:
Population: Participants were not assigned to study arms
Units Other Than Participants: parks
Groups:
- Total: Total of all reporting groups
Arm/Group | Frequent User Arm | Free Physical Activity Classes/Programs | Combined Arm | Control | Total
Number analyzed (Participants) | NA | NA | NA | NA | NA
Number analyzed (parks) | 12 | 12 | 12 | 12 | 48
Age, Categorical [Count of Units; unit: parks] — Age data are not relevant to parks
  parks
    <=18 years | NA — Age is not relevant to parks | NA — Age is not relevant to parks | NA — Age is not relevant to parks | NA — Age is not relevant to parks | NA — Total not calculated because data are not available (NA) in one or more arms.
    Between 18 and 65 years | NA — Age is not relevant to parks | NA — Age is not relevant to parks | NA — Age is not relevant to parks | NA — Age is not relevant to parks | NA — Total not calculated because data are not available (NA) in one or more arms.
    >=65 years | NA — Age is not relevant to parks | NA — Age is not relevant to parks | NA — Age is not relevant to parks | NA — Age is not relevant to parks | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Units; unit: parks] — Gender data are not relevant to parks
  parks
    Female | NA — Gender is not relevant to parks | NA — Gender is not relevant to parks | NA — Gender is not relevant to parks | NA — Gender is not relevant to parks | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — Gender is not relevant to parks | NA — Gender is not relevant to parks | NA — Gender is not relevant to parks | NA — Gender is not relevant to parks | NA — Total not calculated because data are not available (NA) in one or more arms.
park size, [Mean (Full Range); unit: acres] | 6.1 [2.6 to 10.6] | 9.0 [1.9 to 19.2] | 8.0 [1.9 to 25.8] | 10.3 [1.5 to 25.0] | 8.4 [1.5 to 25.8]
population density [Number; unit: people] | 659102 | 583346 | 603596 | 664846 | 2510890

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Park-based Physical Activity
Description: Physical activity was measured in MET-hours (Metabolic equivalents)
Time Frame: difference between baseline and follow-up (1 year)
Population: The unit of analysis was at the level of the park.
Measure: Mean (95% Confidence Interval); unit: Percent change in MET-hours
Units Other Than Participants: Parks
Arm/Group | Frequent User Arm | Free Physical Activity Classes/Programs | Combined Arm | Control
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (Parks) | 12 | 12 | 12 | 12
Percent change in MET-hours | 11.2 [-6.2 to 28.6] | 6.1 [-7.2 to 19.4] | 5.6 [-9.9 to 21.1] | 8.4 [-4.9 to 21.7]
Statistical Analysis 1: Comparison: Frequent User Arm vs Free Physical Activity Classes/Programs vs Combined Arm vs Control; Comparison of change from baseline;; Test type: Superiority — We fitted difference-in-differences (DID) models between the two measurement waves and four study arms. The effect of the intervention was modeled as the wave by study arm interaction. All models used random effects to account for intra-class correlation within each park as well as fixed effects to account for observation times (time of day, weekend versus weekdays); p = .0063, negative binomial distribution — Significance threshold. p=0.05

2. Secondary Outcome: Park Use (% Change)
Description: We will count the number of parks users and compare differences between the number counted at baseline to the number counted at follow-up
Time Frame: baseline versus 1 year
Population: Participants were not assigned to study arms
Measure: Mean (95% Confidence Interval); unit: percentage change in park users
Units Other Than Participants: parks
Arm/Group | Frequent User Arm | Free Physical Activity Classes/Programs | Combined Arm | Control
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (parks) | 12 | 12 | 12 | 12
percentage change in park users | 10 [-9.4 to 29.4] | 4.0 [-10.3 to 18.3] | 6.6 [-11.6 to 24.8] | 9.7 [-2.7 to 22.0]

ADVERSE EVENTS:
Time Frame: Two years
Description: Adverse events occurred if there was any injury associated with our intervention.
Arm/Group | Frequent User Arm | Free Physical Activity Classes/Programs | Combined Arm | Control
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Park observations were snapshot direct observations of aggregated activities. Resident surveys were based on self-reports, subject to reporting biases. The resident sample was a repeated-cross sectional sample rather than a longitudinal cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-10-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT01925404/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT01925404/SAP_001.pdf